CLINICAL TRIAL: NCT01224704
Title: Assessment of Thirst and Role of Water/Electrolytes Homeostasis During Water Deprivation in Obesity
Brief Title: Water Deprivation Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 999911008; 11-DK-N008
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-12-23

CONDITIONS: Obesity
Keywords: Hypertonic Saline Infusion; Water Deprivation; Thirst; Water/Electrolytes Homeostasis; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lean: hypertonic first (Experimental): Lean: Hypertonic solution at day 6 and water deprivation at day 10
  Interventions: Other: Hypertonic saline infusion; Other: Water deprivation
- Lean: water deprivation first (Experimental): Lean: Water deprivation at day 6 and hypertonic solution at day 10
  Interventions: Other: Hypertonic saline infusion; Other: Water deprivation
- Obese: hypertonic first (Experimental): Obese: Hypertonic solution at day 6 and water deprivation at day 10
  Interventions: Other: Hypertonic saline infusion; Other: Water deprivation
- Obese: water deprivation first (Experimental): Obese: Water deprivation at day 6 and hypertonic solution at day 10
  Interventions: Other: Hypertonic saline infusion; Other: Water deprivation

INTERVENTIONS:
Other: Hypertonic saline infusion — Three percent saline (0.1ml/kg of the lean mass/min) will be infused for 120 minutes.
Other: Water deprivation — 24 hour water deprivation

SUMMARY:
Background:

- One area in which obese and lean individuals may be different is how their bodies handle water balance and thirst. Studies done in animals suggest that individuals with greater body fat may tolerate periods without water better than lean animals. Other research has found a link between the ability to tolerate periods without water and increased body weight. Researchers are interested in studying whether the ability to tolerate periods without water and ability to feel thirst might differ in lean versus obese individuals.

Objectives:

- To evaluate the effects of water deprivation and feelings of thirst in lean and obese individuals.

Eligibility:

- Healthy individuals at least 18 years of age who are either lean (body mass index less than 26 kg/m(2)) or obese (body mass index at least 35 kg/m(2)).

Design:

* Participants will be screened with a medical history, physical examination, and blood and urine tests.
* Participants will spend the entire study (13 days) as inpatients at the National Institutes of Health Clinical Center.
* Participants will have the following tests and procedures:
* Body composition assessment (using low-level x-rays) to determine the percentage of fat tissue in the body.
* Oral glucose tolerance test (similar to that often used to diagnose diabetes). Individuals who are suspected to have diabetes will not be allowed to continue with the study.
* High salt infusion test, in which an infusion of saline (salt water) will be given for 2 hours and participants will respond to questions about how hungry and thirsty they feel during the procedure.
* Water deprivation test, in which participants will go for 24 hours without water or food and respond to questions about how hungry and thirsty they feel.
* 24-hour stay in a metabolic chamber to determine how many calories participants burn in a day.
* A series of questionnaires about participants' eating habits, feelings about food, and personal feelings, as well as computer-based tests involving the performance of various tasks.
* Measurement of free-living energy using doubly-labeled water, in which participants will drink a sample of water with extra-heavy atoms of hydrogen and oxygen to evaluate the amount of water in the body.
* 24-hour urine collection.
* Frequent blood samples, urine collection, and fat tissue biopsies during the various study procedures.
* After the end of the 13-day study, participants will return after 1 week for a final urine collection....

DETAILED DESCRIPTION:
Study Description:

The percentage of people with overweight / obesity in the United States has reached very high levels, with 65% of adults over the age of 20 being overweight. Recently, there have been a number of advances in our understanding of the underlying causes of obesity, including greater understanding of both the effects of the environment and effects that are hereditary (i.e., genetic).

One area in which obese versus lean individuals may be different is how their bodies handle water balance and thirst. Studies done in animals suggest that individuals with greater body fat may tolerate periods without water better than lean animals. Thus, at least in animals, others have found a link between ability to tolerate periods without water and increased body weight.

We are studying whether the ability to tolerate periods without water and ability to feel thirst might differ in lean versus obese individuals. To do so, we will ask lean and obese individuals to undergo tests that include a period of approximately 24 hours without drinking any water, and on a separate day a shorter period of an intravenous high salt solution infusion. We will be looking at how the ability to withstand thirst (dehydration), subsequent water intake (rehydration), changes in hormone levels during these periods, and behavioral and physiological responses to thirst and rehydration differ in lean versus obese individuals. We hope that the data gathered from this study will give us more information about important differences in how water balance is regulated in lean versus obese individuals. Understanding these questions may provide new insights into differences between lean and obese individuals.

Objectives:

Primary Objective: to determine if obese versus lean individuals differ in their response (as measured by objective measurement of water intake) to water deprivation and hyperosmolality (dehydration).

Secondary Objective: to determine if during these challenges there are differences in hormonal responses to dehydration and subsequent rehydration, and how these changes are related to adiposity and adipose tissue metabolism.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male.
* Age 18-50 yrs to minimize hormonal influences on thirst perception in aging men.
* BMI<25 kg/m^2 for the lean group and BMI >=35 kg/m^2 for obese group (but weigh less than 350 pounds to accommodate the DXA scanner) for the obese group.
* Healthy, as determined by medical history and physical examination, without the exclusions listed below:

EXCLUSION CRITERIA:

History or Clinical Manifestation of:

* Currently smoking
* Any medications
* Weight <50kg (as the blood withdrawal limit would be exceeded)
* Hemoglobin concentration < 12mg/dl on screening labs
* Type 1 or type 2 diabetes (according to World Health Organization diagnostic criteria (59))
* Endocrine disorders (Cushing's disease, pituitary diseases, hypo- or hyperthyroidism, diabetes insipidus, SIADH)
* Hypertension as diagnosed and treated by an outside physician or by sitting blood pressure measurement, using an appropriate cuff, >140/90 mmHg on two or more occasions
* Fasting triglyceride concentrations >= 500 mg/dl
* Cardiovascular disease, including coronary heart disease, heart failure, arrhythmias and peripheral arterial disease
* Liver disease, including cirrhosis, active hepatitis B or C and AST or ALT >= 3x normal
* Renal disease, as defined by serum creatinine concentrations >= 1.5 mg/dl and / or proteinuria >300 mg/day (200 (micro)g/min)
* Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have been clearly cured or, in the opinion of the investigator, carry an excellent prognosis
* Infectious diseases such as active tuberculosis, HIV (by self report), chronic coccidioidomycoses or other chronic infections
* Alcohol and/or current use of drugs (more than 2 drinks per day and regular use of drugs such as amphetamines, cocaine, heroin, or marijuana)
* Psychiatric conditions or behaviors that would be incompatible with safe and successful participation in this study, including claustrophobia and eating disorders such as anorexia or bulimia nervosa

All subjects will be fully informed of the aim, nature, and risks of the study prior to giving written informed consent. Subjects will also be specifically advised that the results of testing for drug usage will be filed in the medical record and would, therefore, be available as part of this record.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-10-19 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Water intake | End of 24 hour intervention
  Water intake (ml/kg body weight) over the first hour following water deprivation or saline infusion

SECONDARY OUTCOMES:
Hormonal response | During and at the end of intervention
  Vasopressin, apelin, renin-angiotensis system, natriuretic peptides in blood
Thirst rating | During and at the end of interventions
  Thirst is measured by questionnaire using a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marci E Gluck, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Esslinger KA, Jones PJ. Dietary sodium intake and mortality. Nutr Rev. 1998 Oct;56(10):311-3. doi: 10.1111/j.1753-4887.1998.tb01667.x. PMID 9810812
- [Background] Cohen HW, Hailpern SM, Fang J, Alderman MH. Sodium intake and mortality in the NHANES II follow-up study. Am J Med. 2006 Mar;119(3):275.e7-14. doi: 10.1016/j.amjmed.2005.10.042. PMID 16490476
- [Derived] Stinson EJ, Graham AL, Thearle MS, Gluck ME, Krakoff J, Piaggi P. Cognitive dietary restraint, disinhibition, and hunger are associated with 24-h energy expenditure. Int J Obes (Lond). 2019 Jul;43(7):1456-1465. doi: 10.1038/s41366-018-0305-9. Epub 2019 Jan 16. PMID 30651576
- [Derived] Stinson EJ, Krakoff J, Gluck ME. Depressive symptoms and poorer performance on the Stroop Task are associated with weight gain. Physiol Behav. 2018 Mar 15;186:25-30. doi: 10.1016/j.physbeh.2018.01.005. Epub 2018 Jan 9. PMID 29326031